CLINICAL TRIAL: NCT02818192
Title: Improving Renal Complications in Adolescents With Type 2 Diabetes Through REsearch Cohort Study (National iCARE Study)
Acronym: iCARE
Status: Recruiting | Type: Observational
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Brandy Wicklow, Assistant Professor, Pediatrics and Child Health, University of Manitoba
Other Study IDs: B2011:024
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Type 2 Diabetes; Proteinuria; Stress; Nephropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Proteinuria; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, random urine and buffy coat for DNA extraction will be collected at the baseline visit on all recruited patients that consent to biobanking such that future ancillary studies can be performed. Samples will be processed and frozen at -80 °C, and will be stored for up to 25 years with participant consent. Tests that may be run on stored samples include metabolomics, peptidomics, proteomics, and podocyte microparticle analyses should additional funding be obtained. Samples will be collected at each site and frozen. Periodically samples will be sent to the Canadian Biosample Repository at the University of Alberta for long term storage.
Oversight: Data Monitoring Committee: No

SUMMARY:
The overall aim of the project is to elucidate the primary bio-psycho-social (BPS) risk factors for albuminuria in youth with type 2 diabetes (T2D) and the mechanisms by which they cause renal injury. The Study aims include:

1. Characterize the primary BPS risk factors associated with prevalent and progressive albuminuria in youth with T2D.
2. Determine individual, family and community level factors that influence biological and psychological risk factors and behaviors (adherence) that could be modified to protect against prevalent and progressive albuminuria.
3. Determine if systemic and renal inflammation is the common pathway through which BPS risk factors lead to albuminuria in youth with T2D.

Study Hypotheses include:

1. Biological factors (poor glycemic control and systolic ambulatory hypertension), and psychological and social adversity (stress, mental distress and poverty) are significant predictors of prevalent and progressive albuminuria in youth with T2D.
2. Community and family support will be negatively associated with stress, and a lower risk of both prevalent and progressive albuminuria.
3. Systemic and renal inflammation is the common pathway through which BPS risk factors lead to albuminuria in youth with T2D.

DETAILED DESCRIPTION:
The investigators will conduct a case-control study within a two-year, prospective observational cohort study of 500 prevalent cases of T2D diagnosed <18 years of age. The investigators will evaluate the primary BPS risk factors associated with prevalent albuminuria using a principal component analysis (PCA) of associations between primary exposure variables at enrollment. After confirming the relevant BPS factors in the PCA analysis, the investigators will utilize a structural equation modeling approach to confirm the developed model.

ELIGIBILITY:
Inclusion Criteria:

* All youth with T2D that do not meet exclusion criteria are eligible for the study.

Criteria for Diagnosis of T2D:

1. Diagnosis of diabetes will be made according to the Canadian Diabetes Association criteria. There must be 2 abnormal blood glucose tests on different days OR 1 abnormal blood glucose test + symptoms of diabetes:

   * Fasting plasma glucose of > 7.0 mmol/L or
   * Random glucose > 11.1mmol/L or
   * 2 hour glucose > 11.1 mmol/L after a standard oral glucose tolerance test (75g) or
   * Hemoglobin A1c value ≥ 6.5%
2. Distinguishing T2D from type 1 diabetes (T1D) will be based on clinical risk factors including:

   * Presence of overweight/obesity,
   * Other evidence of insulin resistance (acanthosis nigricans)
   * Family history of type 2 diabetes (1st degree relative)
   * Intrauterine exposure to hyperglycemia,
   * Family heritage from a high-risk ethnic group (Indigenous, Hispanic, South Asian, Asian or African descent)
   * Absence of diabetes associated auto-antibodies
   * HNF-1 alpha heterozygote or homozygote

Exclusion Criteria:

1. Diabetes secondary to medication use or surgery
2. Antibodies suggestive of type 1 diabetes
3. Current treatment with oral steroids or immunosuppressive agents as they may interfere with cortisol assessment and inflammatory markers
4. Ever cancer
5. Other chronic illness associated with systemic inflammation (ex. Juvenile rheumatoid arthritis, Crohns disease)
6. Patient and or caregiver unable or unwilling to provide voluntary informed assent/consent

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Prevalent youth 10-18 years of age being treated for T2D at 7 pediatric endocrinology clinics across Canada (Stollery Hospital in Edmonton, Alberta Children's Hospital in Calgary, Children's Hospital of Saskatoon, Children's Hospital of Winnipeg, Children's Hospital of Eastern Ontario in Ottawa, SickKids Hospital in Toronto, and the IWK Health Centre in Halifax)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Persistent Albuminuria | 2 years
  Persistent albuminuria
  Definition:
  1. Albumin:creatine (ACR) > 3.0mg/mmol in at least two urine samples within 6 months at least 1 month apart.
  2. ACR > 3.0mg/mmol with a timed overnight urine or first am urine collection.
Change in albumin excretion over time. | 2 years
  Change in albumin excretion over 2 years. The change in albumin:creatinine ratio, treated as a continuous outcome measure was selected as a valid evaluation of progression of renal injury over time.

SECONDARY OUTCOMES:
Change in estimated glomerular filtration rate (eGFR) over time. | 2 years
  This outcome will be exploratory as significant changes are not expected during a 2-year follow-up period. However, as GFR reflects actual kidney function, this outcome will become increasingly important as chronic kidney disease (CKD) progresses in the cohort over time. GFR will be determined with serum creatinine measurements, utilizing a new eGFR formula for overweight youth, which have been validated utilizing iohexol GFR data from the initial cohort.
  eGFR will be calculated with the iCARE equation. This equation was previously validated for use in the iCARE cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Brandy A Wicklow, MD, MSc, Principal Investigator — University of Manitoba, Children's Hospital Research Institute of Manitoba
Locations (1):
- Children's Hospital Research Institute of Manitoba/University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided
This is a multi-site trial where the use and compilation of individual level data is being discussed amongst the various ethics boards across Canada.

REFERENCES:
- [Result] Dart AB, Wicklow BA, Sellers EA, Dean HJ, Malik S, Walker J, Chateau D, Blydt-Hansen TD, McGavock JM; iCARE investigators. The Improving Renal Complications in Adolescents With Type 2 Diabetes Through the REsearch (iCARE) Cohort Study: rationale and Protocol. Can J Diabetes. 2014 Oct;38(5):349-55. doi: 10.1016/j.jcjd.2014.07.224. PMID 25284698